CLINICAL TRIAL: NCT04685382
Title: Association of Protein Intake With Sarcopenia Among Institutionalized Elderly
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fiastuti Witjaksono, Dr. dr. Fiastuti Witjaksono, MKM, MS, Sp.GK (K), Indonesia University
Other Study IDs: 19-04-0421
Record Dates: First submitted 2020-12-14; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Sarcopenia; Protein Deficiency
Keywords: Protein Intake; Sarcopenia; Institutionalized elderly
MeSH Terms: conditions — Sarcopenia; Protein Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study has purpose to investigated the association of protein intake with sarcopenia in the institutionalized elderly at south tangerang

DETAILED DESCRIPTION:
Data were collected using interview with subjects or with care giver to know the basic characteristic of subjects. Anthropometric measurements were done body weight in kilograms was measured using SECA scale. Body height in meters was predicted by knee height measurement using knee height caliper. Body mass index (BMI) was calculated as weight per height square. Fat free mass was examined using bioelectrical impedance analyzer Tanita type SC-330. Independency was assessed using Barthel index. Protein intake was measured using 2x24 hour food recall and analyzed using a computer program Nutrisurvey 2007, data were compare to Recommended Dietary Allowances established for Indonesian 2018. Handgrip muscle strength was examined using Jamar handgrip dynamometer. Physical performance was measured using Short Physical Performance Battery test. Sarcopenia was diagnosed using Asian Working Group on Sarcopenia.

All data collected were analyzed using Statistical Package for the Social Science (SPSS) version 20 for windows. Nominal data were described using frequency, n (%). Normality of data was tested using Kolmogorov-Smirnov test with normal distribution (p>0.05) described using mean and SD while not normal distribution (p<0.05) described using median and range minimum-maximum. The investigators used Independent T-test analysis to investigate the association.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria were being male or female
2. aged more than 60 years old
3. signed inform consent form and literate with help from companion

Exclusion Criteria:

1. subjects with history of cancer
2. history of upper and lower extremities weakness
3. history of chronic heart failure disease
4. chronic obstructive pulmonary disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited using proportional random sampling method
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Protein intake of the subject | After signing the consent
  to assessed protein intake of the subject using 2x24 hour food recall and analyzed using a computer program Nutrisurvey 2007, data were compare to Recommended Dietary Allowances established for Indonesian 2018
Distribution of sarcopenia subject in the institutionalized elderly | After signing the consent
  to investigate the distribution of sarcopenia subject using Asian Working Group Of Sarcopenia for diagnostic (fat Free Mass, handgrip strength,physical performance) Sarcopenia categorized low muscle mass (fat free mass) and either low muscular strength or low physical performance
Characteristic of fat free mass subject | After signing the consent
  to examine fat free mas of the subject using bioelectrical impedance analyzer Tanita type SC-330 and classified by Asian gender and aged Male : Normal 53,30±4,79 kg Female : Normal 37,96±3,41 kg
Characteristic of handgrip strength subject | After signing the consent
  to assessed handgrip strength of the subject using Jamar handgrip dynamometer, assessment criteria based on the Asian Working Group on Sarcopenia Male : Normal > 26 kg Female : > 18 kg
Characteristic of physical performance subject | After signing the consent
  to examine physical performance (lower extremity strength) using Short Physical Performance Battery test. Classified using Asian Working Group on Sarcopenia Good physical performance score ≥9
Association of protein intake with sarcopenia | immediately after the procedure
  to investigate the association of protein intake with sarcopenia. After protein intake and sarcopenia analysis were completed. The investigators used Independent T-test to analyzed the association protein intake between sarcopenia subject compare to non-sarcopenia subject

SECONDARY OUTCOMES:
Nutritional status of the subjects | After signing the consent
  to investigate nutritional status using anthropometric measurements were done body weight in kilograms was measured using SECA scale. Body height in meters was predicted by knee height measurement using knee height caliper. Body mass index (BMI) was calculated as weight per height square (kg/m2). Nutritional status categorized using WHO Asia Pacific body mass index. Categorized: < 18,5 kg/m2 : underweight 18,5-22,9 kg/m2: normal 23-24,9 kg/m2: overweight >25 kg/m2: obese 1
  ≥30 kg/m2 : obese 2
Barthel index of the subject | After signing the consent
  to know independency of the subject using barthel index scoring
  Scoring:
  Independent : 20 Mild Dependency : 12-19 Moderate Dependency : 9-11 Severe Dependency : 5-8 Total : 0-4 Independent, n (%) Mild Dependency, n (%) Moderate Dependency, n (%) Severe Dependency, n (%)

CONTACTS AND LOCATIONS:
Overall Officials: Fiastuti Witjaksono, Principal Investigator — Department of Nutrition, Faculty of Medicine of Universitas Indonesia
Locations (1):
- Fiastuti Witjaksono, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No